CLINICAL TRIAL: NCT06771531
Title: Cortical Mechanisms and Modulation of Somatosensation in Older Adults With Foot Sole Somatosensory Impairments
Brief Title: Brain Stimulation for Foot-sole Sensation in Older Adults With Foot-sole Somatosensory Deficits
Acronym: BSFS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00044674; K01AG075180 (NIH)
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Somatosensory Function; Balance Control; Mobility
Keywords: brain stimulation; balance and mobility; foot-sole somatosensory function
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tDCS group (Experimental): Participants in this arm will receive the real tDCS intervention.
  Interventions: Device: transcranial direct current stimulation
- sham group (Sham Comparator): Participants in this arm will receive the sham stimulation as control.
  Interventions: Device: active sham stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — tDCS can safely and selectively modulate cortical excitability (specifically neuronal firing likelihood) by transferring weak electrical currents between scalp electrodes. The direct current delivered by any one electrode will not exceed 2.0 mA and the total amount of current from all electrodes will not exceed 4 mA in this study.
  Arms: tDCS group
Device: active sham stimulation — sham stimulation will implement the same protocol of the tDCS intervention; however, only very low-level currents (no more than 0.5 mA) are transferred between the same electrodes used for the tDCS throughout the 20-minute session. This strategy effectively mimics the cutaneous sensations and skin redness induced by creating only micro cortical electric fields.
  Arms: sham group

SUMMARY:
In older adults, diminished sensation of the legs and feet is highly prevalent and causes poor balance and reduced mobility. This type of sensation is not only dependent upon the receptors and nerves in the legs and feet, but also upon a complex central nervous system pathway that includes the cerebral cortex of the brain. This project will use a form of noninvasive brain stimulation called transcranial direct current stimulation (tDCS) to test whether increasing the excitability of the brain networks that process sensory feedback can augment foot sole sensation, balance, and mobility in older adults suffering from mild-to-moderate foot sole sensory impairments.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥65 years.
2. Self-reported feeling of unsteadiness or difficulty when standing and walking.
3. Mild-to-moderate foot-sole somatosensory impairment: the ability to perceive 75g monofilament but inability to perceive 10g monofilament.

Exclusion Criteria:

1. self-reported inability to stand or walk continuously for one minute without personal assistance (canes or walkers allowed);
2. history or presence of foot ulceration, amputation, or deformities;
3. self-reported uncontrolled pain or pain that is associated with mobility disability;
4. uncontrolled diabetes mellitus;
5. hospitalization within the past three months due to acute illness, or as the result of a musculoskeletal injury significantly affecting balance;
6. persistent severe pain of lower extremity when standing or walking;
7. diagnosis of dementia, Parkinson's disease, or stroke that affects balance;
8. unstable medical condition;
9. legal blindness or deafness;
10. uncontrolled hypertension (i.e., systolic BP >180, diastolic BP >100 mm Hg, or prescription of ≥3 anti-hypertensive medications);
11. functionally limiting nephropathy, severe diseases or transplant of the kidney or liver, renal or congestive heart failure;
12. active cancer treatment;
13. balance disorders due to past use of chemotherapy or history of Guillain-Barré syndrome;
14. use of neuro-active or recreational drugs (e.g., sedatives, anti-psychotics), or alcohol abuse, which may affect the brain excitability;
15. contraindications to MRI or tDCS (e.g., personal or family history of seizures or epilepsy, metallic or electric bio-implants, claustrophobia, brain surgery);
16. persistent vertigo;
17. history of Charcot-Marie-Tooth nerve disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
postural sway area when standing with eyes closed on the foam | Before and immediately after intervention
  This metric assesses the degree to which the soft support and cut-off of the vision diminishes the control of standing posture.
Timed Up-and-Go (TUG) time | Before and immediately after intervention
  This metric assesses mobility.
On-target Blood oxygen level dependent (BOLD) signal intensity in response to foot sole stimulation | Before and immediately after intervention
  This metric assesses the degree to which brain cortical regions activated by the walking-related foot-sole stimulation.
Standing vibratory thresholds of each foot sole | Before and immediately after intervention
  This metric assesses the degree to which the foot soles can sense the vibro-tactile stimuli when standing.

SECONDARY OUTCOMES:
Postural sway speed when standing with eyes closed on the foam | Before and immediately after intervention
  This metric assesses the degree to which the soft support and cut-off of the vision diminishes the control of standing posture.
Gait speed of 10m walking test | Before and immediately after intervention
  This metric assesses mobility.

OTHER OUTCOMES:
BOLD signal intensity within other relevant cortical regions in response to foot sole stimulation | Before and immediately after intervention
  This metric assesses the degree to which brain cortical regions activated by the walking-related foot-sole stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebrew SeniorLife, Roslindale, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No